CLINICAL TRIAL: NCT02348060
Title: Autologous Adipose Stromal Vascular Fraction Outcomes in Chronic Obstructive Pulmonary Disease Research Study
Brief Title: Outcomes Data of Adipose Stem Cells to Treat Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: StemGenex (Industry)
Responsible Party: Sponsor
Other Study IDs: SVF01COPD; ASCCOPD-01 (Other: StemGenex)
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the impact that treatment with a cellular concentrate derived from an individual's own fat, known as the stromal vascular fraction (SVF), has on the quality of life of people with chronic obstructive pulmonary disease (COPD). SVF contains multiple cellular components, including stem cells, with both regenerative and anti-inflammatory properties. This therapy has shown promise for ameliorating the symptoms of COPD. This study is designed to evaluate quality of life changes in individuals with COPD for up to 12 months following SVF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with chronic obstructive pulmonary disease (COPD)
* Subjects scheduled for a stem cell/SVF treatment
* Subjects willing and able to sign informed consent
* Subjects willing and able to perform follow-up interviews and surveys

Exclusion Criteria:

* Subjects with additional major health condition/disease diagnoses
* Subjects that are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Overall Quality of Life Over the Course of a 12 Month Period as Measured by the Chronic Respiratory Disease Questionnaire - Self-Administered Individualized (CRQ-SAI) | Baseline, 12 Months
  The change from baseline over the course of 12 months using participants' assessment of their overall quality of life. Mean scores will be used for baseline (day 0) and all interviews up to month 12 (months 1, 3, 6, and 12). Answer options are given as a seven point Likert response scale.

SECONDARY OUTCOMES:
Change from Baseline in Overall Breathing Comfort at Month 12 as Measured by Participants' Responses to the Chronic Respiratory Disease Questionnaire - Self-Administered Individualized (CRQ-SAI) Dyspnea Subscale | Baseline, Month 12
  Participant assessment of breathing comfort from baseline to month 12 using the CRQ-SAI dyspnea subscale.
Change from Baseline in Overall Fatigue at Month 12 as Measured by Participants' Responses to the Chronic Respiratory Disease Questionnaire - Self-Administered Individualized (CRQ-SAI) Fatigue Subscale | Baseline, Month 12
  Participant assessment of fatigue from baseline to month 12 using the CRQ-SAI fatigue subscale.
Change from Baseline in Overall Emotional Function at Month 12 as Measured by Participants' Responses to the Chronic Respiratory Disease Questionnaire - Self-Administered Individualized (CRQ-SAI) Emotional Function Subscale | Baseline, Month 12
  Participant assessment of emotional function from baseline to month 12 using the CRQ-SAI emotional function subscale.
Change from Baseline in Mastery at Month 12 as Measured by Participants' Responses to the Chronic Respiratory Disease Questionnaire - Self-Administered Individualized (CRQ-SAI) Mastery Subscale | Baseline, Month 12
  Participant assessment of mastery (the ability to control feelings of disease-related fear or panic) from baseline to month 12 using the CRQ-SAI mastery subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- StemGenex, San Diego, California, United States